CLINICAL TRIAL: NCT03982940
Title: Physician-Initiated Trial Investigating the BeGraft Peripheral Plus Stent Graft System as Bridging Stent in BEVAR for Complex Aortic Aneurysms
Brief Title: BGP+ Stent as Bridging Stent in BEVAR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marc Bosiers, MD (Other)
Collaborators: Bentley InnoMed GmbH (Industry)
Responsible Party: Sponsor-Investigator, Marc Bosiers, MD, Director, FCRE (Foundation for Cardiovascular Research and Education)
Organization: FCRE (Foundation for Cardiovascular Research and Education) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCRE-190129
Record Dates: First submitted 2019-06-06; First posted 2019-06-12 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Thoracoabdominal Aortic Aneurysm, Without Mention of Rupture
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Intervention Model Description: Application of BeGraft Peripheral Plus (BGP+) Stent Graft System as bridging stent in Branched Endovascular Repair (BEVAR) for complex aortic aneurysms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BGP+ Stent Graft System (Experimental): Application of BeGraft Peripheral Plus (BGP+) Stent Graft System as bridging stent in Branched Endovascular Repair (BEVAR) for complex aortic aneurysms
  Interventions: Device: BGP+ Stent Graft System as bridging stent

INTERVENTIONS:
Device: BGP+ Stent Graft System as bridging stent — BGP+ Stent Graft System as bridging stent

SUMMARY:
The objective of this clinical investigation is to evaluate, in a controlled setting, the safety and performance of the BGP+ balloon expandable covered stent Graft System (Bentley InnoMed, Hechingen, Germany) implanted as bridging stent in BEVAR (branched endovascular aortic repair) for complex aortic aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. Patient eligible for elective repair of TAAA with BEVAR in accordance with the applicable guidelines for vascular interventions (e.g. Aneurysm size 6cm or aneurysm growth of >5mm within 6 months or 1cm within 1 year)
2. Patient is willing to comply with specified follow-up evaluations at the specified times
3. Patient is >55 years old
4. Patient understands the nature of the procedure and provides written informed consent, prior to enrolment in the trial

   • Patient has a projected life-expectancy of at least 12-months
5. Patient needs to have a landing zone in their target vessel of at least 15 mm, and coverage/ wall adaptation of the BGP+ should be obtained for at least 10 mm.
6. The access vessel for introduction of the sheath through which the BGP+ will be advanced should be at least 3mm (it should be able to fit a 8F sheath)
7. No early important division branch from the target vessel with risk of coverage
8. Absence of pre-existing dissection in the target vessels
9. Target vessels (renal arteries, superior mesenteric artery, and celiac trunk) for the BGP+ must have a diameter between 5 and 10 mm
10. Aortic endoprosthesis with inner branches (can be hybrid or branches only)
11. Hybrid aortic endoprosthesis with fenestrations and branches (at least 2 and only the target vessels which are connected by a branch shall be treated with a study device within this study)
12. At least one target vessel is bridged with only one BGP+ (relining allowed)
13. Full compliance with all inclusion criteria/exclusion criteria and all intraoperative criteria

Exclusion Criteria:

1. Previously implanted stent in the target vessel
2. Renal artery with >100° cranial orientation
3. Patients refusing treatment
4. Patients for whom antiplatelet therapy, anticoagulants or thrombolytic drugs are contraindicated
5. Patients with uncorrected bleeding disorders or heparin induced thrombocytopenia
6. Female patient with childbearing potential not taking adequate contraceptives or currently breastfeeding
7. Any planned surgical intervention/procedure within 30 days of the trial procedure
8. Patients with rupture or any patient considered to be hemodynamically unstable at onset of procedure
9. Patient is currently participating in another conflicting investigational drug or device trial that has not completed the entire follow up period.
10. Patients with diffuse distal disease resulting in poor stent outflow
11. Fresh thrombus formation within the last 14 days
12. Patients with known hypersensitivity to the stent material (L605) and/or PTFE
13. Hybrid Approach (endovascular in combination with open surgery)
14. Patients with a connective tissue disorder
15. Patients with mycotic or inflammatory aneurysm
16. Myocardial infarction or stroke within 3 months prior to the procedure
17. Patients with an unstable angina pectoris or heart insufficiency NYHA 3 or 4
18. Patients with ASA classification 5 or higher
19. Contraindications against contrast enhanced angiography (a.e. massive hyperthyroidism)
20. Patients with increased risk of intraoperative rupture
21. Patients with access vessel which are too tortuous, narrow or any kind of reason that would lead to failure of introducing and advancing an introducer sheath

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy endpoint (1) - Technical success | 1 day post-op
  defined as successfully introduction and deployment of the BGP+ balloon expandable covered Stent Graft System implanted as bridging stent in BEVAR
Efficacy endpoint (2) - Bridging stent patency at 12 months | 12 months post-op
  defined as absence of restenosis (≥50% stenosis) or sole target vessel occlusion based on CT angio at 12 months
Safety endpoint - Absence of procedure related complications and bridging stent related endoleaks at 12 months | 12 months post-op
  Absence of procedure related complications and bridging stent related endoleaks at 12 months

SECONDARY OUTCOMES:
Bridging stent patency post-procedure | 1 day post-op, 6- and 24- months post-op
  defined as absence of restenosis (≥50% stenosis) or sole target vessel occlusion based on Duplex Ultrasound or CT Angio
Freedom from bridging stent related endoleaks post-procedure | 1 day post-op, 6- and 24- months post-op
  Freedom from bridging stent related endoleaks post-op, at 6- and 24- months, based on imaging (duplex ultrasound, CT angiography)
Freedom from bridging stent related secondary intervention | 1 day post-op, 6-, 12- and 24- months post-op
  Freedom from bridging stent related secondary intervention
Freedom from type I & III endoleaks post-procedure post-procedure | 1 day post-op, 6-, 12-, and 24- months post-op
  Freedom from type I & III endoleaks post-op and at 6-, 12- and 24- months, based on imaging (duplex ultrasound, CT angiography)
30-day mortality | 30 days post-op
Freedom from stent graft migration | 1 day post-op, 6-, 12 -and 24- months post-op
  defined as freedom from stent graft migration (more than 10 mm)
Freedom from AAA diameter increase | 6-, 12- and 24- months post-op
  defined as more than 5mm increase in maximum diameter measured at 6-, 12- and 24- months as compared to post-op implantation, based on imaging (duplex ultrasound or CT Angiography)
Freedom from aneurysm related secondary endovascular procedures | 1 day post-op, at 6-, 12- and 24- months post-op
  Freedom from aneurysm related secondary endovascular procedures post-op
Freedom from conversion to open surgical repair post-procedure | 1 day post-op, 6-, 12-, 24- months post-op
  Freedom from conversion to open surgical repair post-op and at 6, 12 and 24 months
Freedom from aneurysm related mortality post-procedure | 1 day post-op, 6-, 12-, 24- months post-op
Freedom from aneurysm rupture post-implantation | up to 12- and 24- months post-op
  Freedom from aneurysm rupture within 12- and 24-months post-implantation
Freedom from any major adverse events post-procedural and at 6 and 12 months | 1 day post-op, 6-, 12- and 24- months post-op
Health Related Quality of Life scores | 12- and 24- months post-op
  Health Related Quality of Life scores at 12- and 24 months post implantation

CONTACTS AND LOCATIONS:
Overall Officials: Martin Austermann, PD. Dr., Principal Investigator — Foundation for Cardiovascular Research and Education
Locations (10):
- Germany (10):
  - Prof. Dr. med. Dittmar Böckler - Klinik für Gefäßchirurgie und Endovaskuläre Chirurgie, Heidelberg, Baden-Wurttemberg
  - Prof. Dr. Jost Philipp Schäfer Klinik für Radiologie und Neuroradiologie, Kiel, Schleswig-Holstein
  - Alexander Gombert, Aachen
  - University Hospital Eppendorf, UKE Hamburg, Hamburg
  - University Hospital Leipzig, Leipzig
  - University Hospital LMU Munich, Munich
  - St. Franziskus Hospital, Münster
  - Klinikum Nürnberg Süd, Nuremberg
  - Karin Pfister, Regensburg
  - Hospital Stuttgart, Stuttgart

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: First patient recruited into a study to obtain the indication for a bridging stent in BEVAR procedures — https://interventionalnews.com/bridging-stents-bevar/